CLINICAL TRIAL: NCT00626405
Title: A Randomized Phase II Trial of Temozolomide (TMZ) and Bevacizumab or ABI-007 (ABX)/Carboplatin (CBDCA) and Bevacizumab in Patients With Unresectable Stage IV Malignant Melanoma
Brief Title: Bevacizumab and Temozolomide or Bevacizumab and Paclitaxel Albumin-Stabilized Nanoparticle Formulation and Carboplatin in Treating Patients With Stage IV Malignant Melanoma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCCTG-N0775; NCI-2009-00667 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000587708 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-02-28; First posted 2008-02-29 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Carboplatin; Taxes; Temozolomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive oral temozolomide on days 1-5 and bevacizumab IV over 30-90 minutes on days 1 and 15.
  Interventions: Biological: bevacizumab; Drug: temozolomide
- Arm II (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15, paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1.
  Interventions: Biological: bevacizumab; Drug: carboplatin; Drug: paclitaxel albumin-stabilized nanoparticle formulation

INTERVENTIONS:
Biological: bevacizumab — Given IV over 30-90 minutes
Drug: carboplatin — Given IV over 30 minutes
  Arms: Arm II
Drug: paclitaxel albumin-stabilized nanoparticle formulation — Given IV over 30 minutes
  Arms: Arm II
Drug: temozolomide — Oral temozolomide on days 1-5
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, paclitaxel albumin-stabilized nanoparticle formulation, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether bevacizumab is more effective when given together with temozolomide or paclitaxel albumin-stabilized nanoparticle formulation and carboplatin in killing malignant melanoma cells.

PURPOSE: This randomized phase II trial is studying the side effects of giving temozolomide together with bevacizumab and to see how well it works compared with giving bevacizumab together with paclitaxel albumin-stabilized nanoparticle formulation and carboplatin in treating patients with stage IV malignant melanoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the anti-tumor activity, in terms of the percentage of patients who are treated with these regimens and who are progression-free at 6 months.
* To assess the safety profile of each treatment regimen.

Secondary

* To estimate the response rate in patients treated with these regimens.
* To estimate the distribution of progression-free survival time and overall survival time of patients treated with these regimens.

Tertiary

* To examine the impact of therapy on angiogenesis and immune homeostasis.

OUTLINE: Patients are stratified according to ECOG performance status (0 vs 1) and location of metastatic disease (M1a [skin or subcutaneous tissue or lymph node only] vs M1b [lung] vs M1c [other visceral sites]) and randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral temozolomide on days 1-5 and bevacizumab IV over 30-90 minutes on days 1 and 15. (closed to accrual 8/21/09)
* Arm II: Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15, paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1.

In both arms, treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection periodically for VEGF plasma levels and analysis of changes in immune homeostasis.

Beginning at study entry, patients are followed up every 3 months for 2 years and then every 6 months for up to 3 years.

ELIGIBILITY:
* Histologic confirmed diagnosis of malignant melanoma

  * Stage IV disease
  * Not amenable tosurgery
* Measurable disease with at least one lesion whose longest diameter canbe measured as ≥ 20 mm by CT or MRI scans OR ≥ 10 mm by spiral CT

  * No disease that is measurable by physical examination only
* No brain metastases per MRI or CT
* No radiographically documented invasion of adjacent organs(duodenum, stomach, etc.) or tumor invading major blood vessels
* ECOG performance status 0-1
* Life expectancy ≥ 4 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL (transfusion allowed)
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL (unless Gilbert syndrome)
* AST ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Urine protein:creatinine ratio < 1.0 at screening ORproteinuria < 2+ by urine dipstick or protein ≤ 1 g by 24-hour urine collection
* Negative serum pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Active infection requiring parenteral antibiotics
* Poorly controlled high blood pressure (≥ 150 mm Hg systolic and/or100 mm Hg diastolic) despite treatment
* NYHA class II-IV congestive heart failure
* Serious cardiac arrhythmia requiring medication
* Myocardial infarction or unstable angina within the past 6 months
* Clinically significant peripheral vascular disease
* Deep venous thrombosis or pulmonary embolus within the past year
* Active bleeding or pathological conditions that carry high risk of bleeding (e.g., known esophageal varices)
* Serious, non-healing wound (including wounds healing by secondary intention), ulcer or bone fracture
* Abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within the past 6 months
* History of CNS disease (e.g., primary brain tumor, vascular abnormalities, etc.)
* Clinically significant stroke or TIA within the past 6 months
* Seizures not controlled with standardmedical therapy
* Peripheral neuropathy ≥ grade 2
* History of other malignancy within the past 5 years except basal cell or squamous cell carcinoma of the skin treatable with local resection only or carcinoma in situ of the cervix
* Significant traumatic injury within the past 4 weeks
* History of hypertensive crisis or hypertensive encephalopathy
* Active or recent (≤ 30 days) history of hemoptysis (≥ ½ teaspoon of bright red blood per episode)
* Known hypersensitivity to any of the components of bevacizumab
* Known to be HIV positive
* Current or known history of hepatitis
* Prior adjuvant chemotherapy and/or immunotherapy for this cancer allowed
* No prior treatment with agents disrupting VEGF activity (i.e., bevacizumab,VEGF-trap, anti-VEGFR Mab)
* No ongoing need for full-dose oral or parenteral anticoagulation
* No ongoing anti-platelet treatment other than low-dose aspirin(i.e., aspirin 81 mg daily)
* No other investigational agents within the past 4 weeks
* No major surgical procedure or open biopsy within the past 4 weeks
* No fine needle aspirations or core biopsies within the past 7 days
* No prior chemotherapy in the metastatic setting
* No prior treatment with sunitinib malate or sorafenib
* No prior treatment with any taxane-based chemotherapy
* Patients who have had > 25% of their functional bone marrow irradiated are not eligible for this trial
* No adjuvant radiation therapy within the past 4 weeks
* More than 2 weeks since prior and no concurrent palliative radiation therapy
* No concurrent major surgical procedure
* No concurrent participation in another clinical study for procedures or agents that treat the same primary study malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, MD, PhD, Study Chair — Mayo Clinic
Locations (259):
- United States (259):
  - Providence Cancer Center, Anchorage, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Kottschade LA, Suman VJ, Perez DG, McWilliams RR, Kaur JS, Amatruda TT 3rd, Geoffroy FJ, Gross HM, Cohen PA, Jaslowski AJ, Kosel ML, Markovic SN. A randomized phase 2 study of temozolomide and bevacizumab or nab-paclitaxel, carboplatin, and bevacizumab in patients with unresectable stage IV melanoma : a North Central Cancer Treatment Group study, N0775. Cancer. 2013 Feb 1;119(3):586-92. doi: 10.1002/cncr.27760. Epub 2012 Aug 22. PMID 22915053

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients receive oral temozolomide on days 1-5 and bevacizumab IV over 30-90 minutes on days 1 and 15.> > bevacizumab: Given IV over 30-90 minutes>
  > temozolomide: Oral temozolomide on days 1-5
- Arm II: Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15, paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1.>
  > bevacizumab: Given IV over 30-90 minutes>
  > carboplatin: Given IV over 30 minutes>
  > paclitaxel albumin-stabilized nanoparticle formulation: Given IV over 30 minutes
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 43 | 52
Completed | 42 | 51
Not Completed | 1 | 1
Not completed — Deemed Ineligible | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients who began treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 42 | 51 | 93
Age, Continuous [Median (Full Range); unit: Years] | 57 [25 to 82] | 57 [22 to 83] | 57 [22 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 24 | 29 | 53

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months
Description: The primary endpoint is the 6 month post registration Progression-free survival (PFS) rate. Progression-free survival time is defined as the time from registration to documentation of disease progression using the RECIST criteria. Patients who died without documentation of disease progression will be considered to have progressed at death unless there is sufficient documented evidence to conclude no progression occurred prior to death. All patients, who meet the eligibility criteria, sign a consent form, and start treatment will be included in the evaluation of the 6 month PFS rate.
Time Frame: at 6 months
Population: The first 41 eligible patients randomized to each treatment arm.
Measure: Number (90% Confidence Interval); unit: % of patients alive and progression free
Groups:
- Arm I: Patients receive oral temozolomide on days 1-5 and bevacizumab IV over 30-90 minutes on days 1 and 15.
  >
  > bevacizumab: Given IV over 30-90 minutes
  >
  > temozolomide: Oral temozolomide on days 1-5
- Arm II: Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15, paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1.
  >
  > bevacizumab: Given IV over 30-90 minutes
  >
  > carboplatin: Given IV over 30 minutes
  >
  > paclitaxel albumin-stabilized nanoparticle formulation: Given IV over 30 minutes
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 41 | 41
% of patients alive and progression free | 32.8 [21.1 to 51.2] | 56.1 [44.7 to 70.4]

2. Secondary Outcome: Tumor Response Rate, Calculated as a Percentage Along With it's 95% Confidence Interval
Description: A confirmed tumor response is defined to be a Complete Response or Partial Response noted
  > as the objective status on 2 consecutive evaluations at least 8
  > weeks apart. The proportion of tumor responses will be
  > estimated by the number of confirmed tumor responses divided
  > by the total number of evaluable patients.
  > Complete Response (CR): Disappearance of all target lesions
  > Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
  > Progression (PD): At least a 20% increase in the sum of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  > Stable Disease (SD): Neither sufficient shrinkage to Qualify for PR nor sufficient increase to Qualify for PD taking as reference the smallest sum LD. responses will be calculated assuming that the number of
  > confirmed tumor responses follows a binomial distribution.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with response
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 42 | 51
percentage of patients with response | 23.8 [12.1 to 39.5] | 33.3 [20.8 to 47.9]

3. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 42 | 51
Months | 12.3 [9.3 to 15.3] | 13.9 [9.8 to 15.5]

ADVERSE EVENTS:
Time Frame: Until treatment discontinuation
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 7/43 | 18/51
Other Adverse Events (participants affected / at risk) | 43/43 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=43) | Arm II (N=51)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2) | 5 (5)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 7 (7)
Platelet count decreased (Investigations) | 3 (3) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=43) | Arm II (N=51)
Hemoglobin decreased (Blood and lymphatic system disorders) | 27 (79) | 46 (279)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (8)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 3 (7)
Constipation (Gastrointestinal disorders) | 2 (3) | 6 (10)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 2 (2)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 2 (4) | 4 (9)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (9)
Nausea (Gastrointestinal disorders) | 32 (130) | 32 (94)
Oral cavity fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 20 (42) | 15 (37)
Disease progression (General disorders) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 42 (207) | 48 (254)
Fever (General disorders) | 9 (10) | 8 (8)
Hypersensitivity (Immune system disorders) | 3 (5) | 5 (7)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 15 (45) | 38 (191)
Lymphocyte count decreased (Investigations) | 0 (0) | 4 (11)
Neutrophil count decreased (Investigations) | 7 (8) | 36 (159)
Platelet count decreased (Investigations) | 17 (64) | 30 (145)
Weight loss (Investigations) | 0 (0) | 5 (10)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 7 (13)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 3 (6)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 17 (69) | 20 (74)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (66) | 18 (54)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (4)
Acoustic nerve disorder NOS (Nervous system disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 3 (14)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (5)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (16) | 24 (85)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (2)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Taste alteration (Nervous system disorders) | 0 (0) | 2 (7)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 14 (29) | 19 (73)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 8 (20) | 15 (41)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (11)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (19)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 23 (62) | 18 (59)
Thrombosis (Vascular disorders) | 3 (4) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes